CLINICAL TRIAL: NCT01335659
Title: Relationship Between Fractional Flow Reserve and Coronary Angiography/Intravascular Ultrasound Parameters in Ostial Lesions: Major Coronary Ostial Lesions Versus Side Branch Ostial Lesions
Brief Title: Main Branch Versus Side Branch Ostial Lesion
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Bon-Kwon Koo / Professor, Seoul National University hospital
Other Study IDs: Bif_3
Record Dates: First submitted 2011-04-07; First posted 2011-04-14 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Stenosis
Keywords: FFR; IVUS; QCA
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ostial lesion: ostial lesion will be evaluated by IVUS and FFR
  Interventions: Device: Fractional flow reserve; Device: IVUS

INTERVENTIONS:
Device: Fractional flow reserve — Fractional flow reserve measured by pressure wire
  Other Names: Radi Pressure Wire(Radi Medical Systems, Uppsala, Sweden)
Device: IVUS — intravascular ultrasound
  :IVUS was performed in a standard fashion using an automated motorized pullback system (0.5mm/s) with commercially available imaging catheter
  Other Names: iLab® Ultrasound Imaging System(Boston Scientific/SCIMED, Minneapolis, MN, USA)

SUMMARY:
The investigators studied the relations between coronary angiography (CAG), intravascular ultrasound (IVUS) and fractional flow reserve (FFR) in coronary ostial lesions.

DETAILED DESCRIPTION:
Angiographic evaluation for ostial lesions is reported to be inaccurate in the assessment of the functional and clinical significance of a lesion. The investigators studied the relations between coronary angiography (CAG), intravascular ultrasound (IVUS) and fractional flow reserve (FFR) in coronary ostial lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-85
* Presence of at least one obstructive coronary artery stenosis at coronary ostium as defined by:
* Previous catheterization with any coronary ostium lesion 50% or greater
* Ability and Willingness to provide informed consent
* Ability and Willingness to perform required follow up procedures

Exclusion Criteria:

* History of coronary artery bypass graft surgery
* left main coronary ostial lesion
* significant stenosis at proximal or distal part of coronary ostium lesion
* ostial lesion related to infarcton
* Creatinine>1.6 mg/dL or GFR<30 pre-procedure per institutional standards
* Ejection fraction lower than 40%
* Known Pregnancy
* Arrhythmia
* Contrast agent allergy that cannot be adequately premedicated
* Patient not a candidate for IVUS and FFR
* Inability or unwillingness to provide informed consent
* Inability or unwillingness to perform required follow up procedures

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: from september 2009 to january 2011 patient who are undergone coronary angiography,IVUS and FFR for the evaluation of coronary artery disease at SNUH
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
lumen area | 1 day
  lumen area at ostial lesion

SECONDARY OUTCOMES:
angiographic stenosis, % plaque area | 1 day
  angiographic and intravascular ultrasound parameters at ostial lesions of each major branch and side branch.

CONTACTS AND LOCATIONS:
Overall Officials: Bon-kwon Koo, MD/PhD, Study Director — Seoul National University Hospital

REFERENCES:
- [Derived] Koh JS, Koo BK, Kim JH, Yang HM, Park KW, Kang HJ, Kim HS, Oh BH, Park YB. Relationship between fractional flow reserve and angiographic and intravascular ultrasound parameters in ostial lesions: major epicardial vessel versus side branch ostial lesions. JACC Cardiovasc Interv. 2012 Apr;5(4):409-15. doi: 10.1016/j.jcin.2012.01.013. PMID 22516397